CLINICAL TRIAL: NCT02298153
Title: A Phase 1 Study of Atezolizumab in Combination With Epacadostat in Subjects With Previously Treated Stage IIIB or Stage IV Non-Small Cell Lung Cancer and Previously Treated Stage IV Urothelial Carcinoma (ECHO-110)
Brief Title: A Study of Atezolizumab (MPDL3280A) in Combination With Epacadostat (INCB024360) in Subjects With Previously Treated Stage IIIB or Stage IV Non-Small Cell Lung Cancer and Previously Treated Stage IV Urothelial Carcinoma (ECHO-110)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention.
Sponsor: Incyte Corporation (Industry)
Collaborators: Hoffmann-La Roche (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 24360-110 / ECHO-110
Record Dates: First submitted 2014-10-31; First posted 2014-11-21 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: NSCLC (Non-small Cell Lung Carcinoma); UC (Urothelial Cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; epacadostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- atezolizumab (MPDL3280A) + epacadostat (INCB024360) (Experimental): atezolizumab (MPDL3280A) 1200 mg given every 3 weeks + epacadostat (INCB024360) 25 mg BID as starting dose, followed by dose escalations until MTD or PAD is identified
  Interventions: Drug: atezolizumab; Drug: epacadostat

INTERVENTIONS:
Drug: atezolizumab — atezolizumab: administered intravenously (IV) every three weeks (q3w)
  Other Names: MPDL3280A
Drug: epacadostat — epacadostat: Oral daily dosing
  Other Names: INCB024360

SUMMARY:
This study will evaluate the safety and tolerability of epacadostat (INCB024360) administered in combination with atezolizumab (MPDL3280A) in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) that have been previously treated with platinum-based chemotherapy and Stage IV urothelial carcinoma who have failed a platinum-based chemotherapy regimen. The study will be conducted in two phases. The dose escalation phase will utilize a 3 + 3 design to identify the maximum tolerated dose (MTD) or a Pharmacologically Active Dose (PAD) of the combination. This will be followed by a dose expansion phase, which will be comprised of three cohorts. Expansion Cohorts 1 & 2 will further evaluate the safety, tolerability, efficacy, pharmacokinetics (PK), and pharmacodynamics at the dose identified in phase one. Expansion Cohort 3 will evaluate the change in biomarker expression following treatment with epacadostat as monotherapy followed by epacadostat and atezolizumab administered in combination.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, age 18 years or older
* Histologically or cytologically confirmed NSCLC
* Stage IIIB or Stage IV NSCLC who are not candidates for multimodality treatment and have received at least 1 line of standard platinum-based therapy:

  * Prior systemic regimens must include at least 2 cycles of a platinum-based therapy and may include platinum therapy used as a radiosensitizer. Maintenance chemotherapy is allowed.
  * Tumors with driver mutations (epidermal growth factor receptor mutation positive or anaplastic lymphoma kinase fusion oncogene positive) should have had disease progression or been intolerant to the standard tyrosine-kinase inhibitor (TKI), and should include a second line TKI where such therapy is available and indicated.
  * Subjects initially treated with a platinum regimen for Stage IIIB disease who later develop metastatic disease and are re-treated with a platinum regimen are allowed.
* Histologically or cytologically confirmed urothelial carcinoma.
* Stage IV locally advanced or metastatic urothelial carcinoma with disease progression during or following platinum-containing chemotherapy or had disease progression within 12 months of neoadjuvant or adjuvant treatment with platinum-containing chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
* Presence of measurable disease per RECIST v1.1
* Availability of an adequate archival tumor specimen or willingness to undergo a pretreatment tumor biopsy.
* Subjects enrolled in Expansion Cohort 3 must be willing to have 2 on-treatment tumor biopsies.
* For males and females of child-bearing potential, willingness to use adequate birth control through 90 days after the last dose of epacadostat or atezolizumab.

Exclusion Criteria:

* Laboratory and medical history parameters not within protocol-defined range.
* Current treatment with an investigational study drug or immunological-based agent for any reason, or receipt of anticancer medication within 21 days or 5 half-lives (whichever is longer) before first dose.
* Prior treatment with immune checkpoint inhibitors (eg, anti-CTLA-4, anti-PD-1, anti-PD-L1, and any other antibody or drug specifically targeting T-cell co-stimulation) or an IDO inhibitor.
* Prior monoclonal antibody within 4 weeks before study Day 1, or has not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Has an active or inactive autoimmune process.
* Has a history of pneumonitis or idiopathic pulmonary fibrosis, or evidence of interstitial lung disease.
* Prior radiotherapy within 2 weeks of therapy; Must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
* Untreated central nervous system (CNS) metastases or CNS metastases that have progressed after completion of radiotherapy.
* Use of systemic corticosteroids ≤ 2 weeks before Cycle 1 Day 1.
* Currently pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Continuously for duration of study participation and up to 42 days after the last dose [approximately 8 months
Incidence of dose-limiting toxicities (DLTs) | 21 days following the first administration of atezolizumab and epacadostat

SECONDARY OUTCOMES:
Objective response rate (ORR) | Measured every 6 weeks for duration of study participation [approximately 8 months]
  ORR determined by radiographic disease assessments per modified RECIST v1.1
Durability of response | Measured every 6 weeks for duration of study participation [approximately 8 months]
  Time from the earliest date of disease response until earliest date of disease progression based on modified RECIST v1.1
Progression-free survival | Measured every 6 weeks for duration of study participation [approximately 8 months]
  Time from date of enrollment until the earliest date of disease progression per modified RECIST v1.1 or death due to any cause, whichever is earlier.
Duration of disease control | Measured every 6 weeks for duration of study participation [approximately 8 months]
  Time from first dose until report of disease progression for subjects who reported stable disease or better based on modified Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Hiroomi Tada, MD, Study Director — Incyte Corporation
Locations (6):
- United States (6):
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - Yale University, New Haven, Connecticut
  - Harvard-Mass General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Washington, Seattle, Washington